CLINICAL TRIAL: NCT01742078
Title: A Single-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY2541546 in Healthy Postmenopausal Women
Brief Title: A Study of LY2541546 in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 11952; I2M-MC-GSDA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: Postmenopausal females; Volunteers
MeSH Terms: interventions — blosozumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- 7.5 mg LY2541546 - IV (Experimental): Single dose of 7.5 mg LY2541546 administered intravenously (IV)
  Interventions: Drug: LY2541546 - IV
- 25 mg LY2541546 - IV (Experimental): Single dose of 25 mg LY2541546 administered IV
  Interventions: Drug: LY2541546 - IV
- 75 mg LY2541546 - IV (Experimental): Single dose of 75 mg LY2541546 administered IV
  Interventions: Drug: LY2541546 - IV
- 225 mg LY2541546 - IV (Experimental): Single dose of 225 mg LY2541546 administered IV
  Interventions: Drug: LY2541546 - IV
- 750 mg LY2541546 - IV (Experimental): Single dose of 750 mg LY2541546 administered IV
  Interventions: Drug: LY2541546 - IV
- 150 mg LY2541546 - SC (Experimental): Single dose of 150 mg LY2541546 administered subcutaneous (SC)
  Interventions: Drug: LY2541546 - SC
- Placebo (Placebo Comparator): Single dose of placebo administered IV or SC
  Interventions: Drug: Placebo
- 225 mg LY2541546 - IV, OL (Experimental): Single dose of 225 mg LY2541546 administered IV, open label (OL)
  Interventions: Drug: LY2541546 - IV
- 750 mg LY2541546 - IV, OL (Experimental): Single dose of 750 mg LY2541546 administered IV, OL
  Interventions: Drug: LY2541546 - IV

INTERVENTIONS:
Drug: LY2541546 - IV — Administered IV
  Other Names: Blosozumab
  Arms: 225 mg LY2541546 - IV; 225 mg LY2541546 - IV, OL; 25 mg LY2541546 - IV; 7.5 mg LY2541546 - IV; 75 mg LY2541546 - IV; 750 mg LY2541546 - IV; 750 mg LY2541546 - IV, OL
Drug: LY2541546 - SC — Administered SC
  Arms: 150 mg LY2541546 - SC
Drug: Placebo — Administered IV or SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if a single dose of LY2541546 has any side effects on the body and to determine how long and how much LY2541546 stays in the bloodstream of the body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal females, as determined by medical history and physical examination
* Body mass index (BMI) at screening between 19.0 and 32.0 kilograms per square meter (kg/m^2), inclusive
* Acceptable Clinical laboratory test results, blood pressure and heart rate
* Have given written informed consent
* Additional Inclusion Criterion for Participants in Open Label Groups: Are currently taking or recently discontinued (not more than 3 months prior to study randomization) alendronate and have taken alendronate for at least 12 of the last 18 months

Exclusion Criteria:

* Within 30 days of the initial dose of study drug, have received treatment with a drug that has not received regulatory approval for any indication
* Known allergies to LY2541546, its constituents, or related compounds
* Persons who have previously participated in this study
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders
* History of or high risk for adverse outcome from bleeding, for example, transient ischemic attacks, cerebrovascular attacks, and ulcer disease
* Paget's disease, parathyroid disease, or thyroid disease
* Fracture of a long bone within 12 weeks of screening
* Regular use of known drugs of abuse and/or positive findings on urinary drug screening
* Evidence of human immunodeficiency virus (HIV), hepatitis C, hepatitis B and/or positive for anti-HIV antibodies, hepatitis C antibody, or hepatitis B surface antigen
* Current use of therapies for osteoporosis or use of hormone replacement therapy (HRT) within the previous 12 months
* Blood donation within the last month
* Participants who have an average weekly alcohol intake that exceeds 14 units per week
* Cigarette consumption of more than 10 cigarettes per day, or are unable or unwilling to refrain from nicotine during Clinical Research Unit (CRU) confinement

Additional Exclusion Criterion for Participants in Double Blind Groups Only

* Have received bisphosphonates during the previous 24 months.

Additional Exclusion Criterion for Participants in Open Label Groups

* Have received intravenous bisphosphonates within the previous 18 months

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 7.5 mg LY2541546 - IV | 25 mg LY2541546 - IV | 75 mg LY2541546 - IV | 225 mg LY2541546 - IV | 750 mg LY2541546 - IV | 150 mg LY2541546 - SC | 225 mg LY2541546 - IV, OL | 750 mg LY2541546 - IV, OL | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12
RECEIVED STUDY DRUG | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12
Completed | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received study drug.
Groups:
- 7.5 mg LY2541546 - IV: Participants received 7.5 mg LY2541546 IV
- 25 mg LY2541546 - IV: Participants received25 mg LY2541546 IV
- 75 mg LY2541546 - IV: Participants received 75 mg LY2541546 IV
- 225 mg LY2541546 - IV: Participants received225 mg LY541546 IV
- 750 mg LY2541546 - IV: Participants received750 mg LY2541546 IV
- 150 mg LY2541546 - SC: Participants received 150 mg LY2541546 subcutaneously (SC)
- 225 mg LY2541546 - IV, OL: Participants received 225 mg LY2541546 IV. Open label(OL)
- 750 mg LY2541546 - IV, OL: Participants received 750 mg LY2541546 IV, OL
- Placebo: Participants single dose of placebo administered IV or SC
- Total: Total of all reporting groups
Arm/Group | 7.5 mg LY2541546 - IV | 25 mg LY2541546 - IV | 75 mg LY2541546 - IV | 225 mg LY2541546 - IV | 750 mg LY2541546 - IV | 150 mg LY2541546 - SC | 225 mg LY2541546 - IV, OL | 750 mg LY2541546 - IV, OL | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (3.7) | 56.3 (4.6) | 60.0 (5.3) | 53.6 (4.6) | 59.0 (5.7) | 58.5 (4.5) | 59.7 (6.7) | 64.2 (5.9) | 57.1 (5.2) | 57.9 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 60
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5 | 5 | 6 | 5 | 5 | 6 | 6 | 6 | 11 | 55
  African | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Native American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  West Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: An SAE is any AE from this study that results in one of the following outcomes:
  * death
  * initial or prolonged inpatient hospitalization
  * a life-threatening experience (that is, immediate risk of dying)
  * persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * or is considered significant by the investigator for any other reason.
Time Frame: Day 1 through Day 85
Population: All participants who received study drug.
Measure: Number; unit: participants
Arm/Group | 7.5 mg LY2541546 - IV | 25 mg LY2541546 - IV | 75 mg LY2541546 - IV | 225 mg LY2541546 - IV | 750 mg LY2541546 - IV | 150 mg LY2541546 - SC | Placebo | 225 mg LY2541546 - IV, OL | 750 mg LY2541546 - IV, OL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve Versus Time Curve From Time Zero to Infinity (AUC0-∞) of LY2541546
Time Frame: Day 1: Predose,30 minutes,45 mintues,1 hour (hr), 1.5 hr, 3 hr, 6 hr, 12 hr Postdose; Day (D) 3,D5 ,D8, D11, D15, D29, D43, D57, D71,D85: anytime
Population: All participants who received study drug and had sufficient evaluable results for PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomol*hr/mL
Arm/Group | 7.5 mg LY2541546 - IV | 25 mg LY2541546 - IV | 75 mg LY2541546 - IV | 225 mg LY2541546 - IV | 750 mg LY2541546 - IV | 150 mg LY2541546 - SC | 225 mg LY2541546 - IV, OL | 750 mg LY2541546 - IV, OL
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6
picomol*hr/mL | 411 (51) | 2540 (22) | 16400 (16) | 86600 (14) | 390000 (14) | 9150 (40) | 94500 (10) | 507000 (14)

3. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline in Lumbar Spine Bone Mineral Density (BMD)
Description: A BMD test measures the amount of mineral (such as calcium) in a defined area of bone in grams per square centimeter (g/cm²) and is calculate by dexascan.
Time Frame: Baseline (predose), Day 29 anytime, Day 85 anytime
Population: All participants who received study drug and had evaluable results at the analyzed time points.
Measure: Least Squares Mean (90% Confidence Interval); unit: gram per square centimeter (g/cm^2)
Arm/Group | 7.5 mg LY2541546 - IV | 25 mg LY2541546 - IV | 75 mg LY2541546 - IV | 225 mg LY2541546 - IV | 750 mg LY2541546 - IV | 150 mg LY2541546 - SC | Placebo | 225 mg LY2541546 - IV, OL | 750 mg LY2541546 - IV, OL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6
gram per square centimeter (g/cm^2)
  Day 29: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 11 | 6 | 6
  Day 29 | 0.01 [-0.01 to 0.02] | -0.01 [-0.03 to 0.01] | 0.01 [-0.00 to 0.02] | 0.01 [-0.00 to 0.03] | 0.00 [-0.01 to 0.02] | 0.00 [-0.01 to 0.01] | -0.00 [-0.01 to 0.01] | 0.01 [-0.00 to 0.03] | -0.00 [-0.02 to 0.01]
  Day 85 | -0.00 [-0.02 to 0.01] | -0.01 [-0.02 to 0.01] | 0.01 [-0.00 to 0.03] | 0.02 [0.00 to 0.03] | 0.03 [0.02 to 0.05] | 0.01 [-0.00 to 0.02] | -0.00 [-0.02 to 0.01] | 0.01 [-0.01 to 0.02] | 0.02 [0.00 to 0.03]

4. Secondary Outcome: Pharmacodynamics (PD): Percent Change From Baseline in N-terminal Propeptide of Procollagen Type 1 (P1NP)
Description: N-terminal propeptide of procollagen type 1 (P1NP) is a main bone formation marker. An increase of P1NP in serum reflects elevated anabolic activities of the bone. Percentage change in P1NP from baseline to post baseline time points was analyzed using the repeated-measures model.
Time Frame: Baseline (predose), Day 29 anytime, Day 85 anytime
Population: All participants who received study drug and had evaluable results at the analyzed timepoints.
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage of change from baseline
Arm/Group | 7.5 mg LY2541546 - IV | 25 mg LY2541546 - IV | 75 mg LY2541546 - IV | 225 mg LY2541546 - IV | 750 mg LY2541546 - IV | 150 mg LY2541546 - SC | Placebo | 225 mg LY2541546 - IV, OL | 750 mg LY2541546 - IV, OL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6
percentage of change from baseline
  Day 29: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 11 | 6 | 6
  Day 29 | 9.36 [-38.79 to 57.52] | 44.00 [-4.15 to 92.16] | 24.86 [-23.30 to 73.01] | 47.54 [-2.50 to 97.59] | 224.16 [176.00 to 272.32] | 31.42 [-16.74 to 79.57] | 6.18 [-28.37 to 40.73] | 106.76 [58.60 to 154.91] | 334.52 [286.36 to 382.68]
  Day 85 | 9.28 [-22.36 to 40.93] | 25.77 [-5.88 to 57.42] | 14.27 [-17.38 to 45.92] | 24.07 [-7.58 to 55.72] | 33.84 [2.20 to 65.49] | 19.24 [-12.41 to 50.89] | 9.86 [-12.52 to 32.24] | 33.59 [1.95 to 65.24] | 23.98 [-7.67 to 55.62]

5. Secondary Outcome: Immunogenicity: The Number of Participants With Anti-LY2541546 Antibodies
Description: A validated assay designed to perform in the presence of LY2541546 was used for to assess development of antibodies.
Time Frame: Day 1: Predose, Day 29 anytime, Day 85 anytime
Population: All participants who received study drug and had evaluable results at the analyzed time points.
Measure: Count of Participants; unit: Participants
Arm/Group | 7.5 mg LY2541546 - IV | 25 mg LY2541546 - IV | 75 mg LY2541546 - IV | 225 mg LY2541546 - IV | 750 mg LY2541546 - IV | 150 mg LY2541546 - SC | Placebo | 225 mg LY2541546 - IV, OL | 750 mg LY2541546 - IV, OL
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6
Participants
  Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 29 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Day 85 | 0 | 0 | 1 | 4 | 1 | 2 | 0 | 0 | 2

ADVERSE EVENTS:
Arm/Group | 7.5 mg LY2541546 - IV | 25 mg LY2541546 - IV | 75 mg LY2541546 - IV | 225 mg LY2541546 - IV | 750 mg LY2541546 - IV | 150 mg LY2541546 - SC | Placebo | 225 mg LY2541546 - IV, OL | 750 mg LY2541546 - IV, OL
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 4/6 | 4/6 | 4/6 | 5/6 | 7/12 | 6/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7.5 mg LY2541546 - IV (N=6) | 25 mg LY2541546 - IV (N=6) | 75 mg LY2541546 - IV (N=6) | 225 mg LY2541546 - IV (N=6) | 750 mg LY2541546 - IV (N=6) | 150 mg LY2541546 - SC (N=6) | Placebo (N=12) | 225 mg LY2541546 - IV, OL (N=6) | 750 mg LY2541546 - IV, OL (N=6)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual disturbance (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days